CLINICAL TRIAL: NCT07037680
Title: Efficiency and Safety of Radiotherapy Combined With Anlotinib in Locally Advanced Non-small Cell Lung Cancer Patients Intolerable to Concurrent Chemoradiotherapy: A Phase II Single-arm Trial
Brief Title: Radiotherapy Plus Anlotinib in LA-NSCLC Intolerable to cCRT
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: JIANYANG WANG (Other)
Responsible Party: Sponsor-Investigator, JIANYANG WANG, Principal Investigator, Cancer Institute and Hospital, Chinese Academy of Medical Sciences
Organization: Cancer Institute and Hospital, Chinese Academy of Medical Sciences (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCC2827
Record Dates: First submitted 2025-05-28; First posted 2025-06-25 (Actual); Last update posted 2025-07-09 (Actual); Status verified 2025-07

CONDITIONS: Locally Advanced Non-Small Cell Lung Cancer; Thoracic Radiotherapy; Safety
Keywords: thoracic radiotherapy; non-small cell lung carcinoma; locally advanced; safety; Anlotinib
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — anlotinib

STUDY DESIGN:
Intervention Model Description: A phase II randomized trial (registered in Clinical Trials.gov as NCT05888402) of unresectable stage III NSCLC patients undergone definitive concurrent chemoradiotherapy was prespecified to compare the 2-year PFS difference with that of current trial.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Radiotherapy plus Anlotinib (Experimental): Radiotherapy plus anlotinib in LA-NSCLC intolerable to cCRT
  Interventions: Drug: Anlotinib

INTERVENTIONS:
Drug: Anlotinib — For patients treated with conventional Intensity-Modulated Radiation Therapy (IMRT), the median prescribed dose was 60 Gy/30 fractions (range: 50.0-70.0 Gy, in 25-35 fractions) (median BED10 72 Gy, range: 60-84 Gy) to the planning target volume (PTV). As for patients with IMRT-based simultaneously integrated boost (SIB), the median prescribed dose was 59.92 Gy/28 fractions (range: 50.0-70.0 Gy, in 25-33 fractions) (median BED10 72.74 Gy, range: 60-84 Gy) to the planning gross tumor volume (PGTV), and 50.4 Gy/28 fractions (range: 45-59.4 Gy, in 25-33 fractions) (median BED10 59.47 Gy, range: 53.1-70.1 Gy) to the PTV. It should be noted that the PTV in the SIB group contains the PGTV.
  Anlotinib was administered orally concurrently with the first day of radiotherapy, at a dose of 12 mg for a maximum of three cycles. Each cycle was defined as 2 weeks on-treatment followed by 1 week off-treatment. If intolerance occurs, the dose may be reduced to 8-10 mg/day or stopped.

SUMMARY:
Concurrent chemoradiotherapy (cCRT) is the standard treatment for patients with negative epidermal growth factor receptor (EGFR)-mutated unresectable locally advanced non-small cell lung cancer (LA-NSCLC). However, parts of patients only receive sequential chemoradiotherapy (sCRT) due to various reasons. This phase II study aimed to improve the outcomes of patients receiving sCRT by combining anti-angiogenesis therapy (Anlotinib) during radiotherapy course.We hypothesize that the combination of radiotherapy with anlotinib could improve the 2-year PFS rate from 35% with sCRT to 50. The accrual target was 44 patients.

ELIGIBILITY:
Patients with histologically or cytologically confirmed negative EGFR (including EGFR exon 19 deletion or L858R mutations) or ALK/ROS1-mutated locally advanced unresectable NSCLC were screened.

Inclusion Criteria:

1. ≥18 years old with no restrictions on sex;
2. Peripheral tumor, or central lung cancer with non-squamous tissue or a mixed tissue with less than 50% squamous carcinoma;
3. Eastern cooperative oncology group (ECOG) score ≤2 was required;
4. Received systemic chemotherapy or combined chemotherapy and immumitherapy for ≥ 4 weeks without progression;
5. .No cavity inside the tumor, and located ≥ 1 cm of the main pulmonary artery trunk;
6. No symptoms of hemoptysis;
7. Adequate hepatic and renal functions with a negative urine protein;
8. Expected survival of more than 6 months.

Exclusion Criteria:

1. currently receiving treatment for malignancies at other sites, except for curable non-melanoma skin cancer and cervical carcinoma in situ;
2. previous malignancy within five years;
3. thoracic radiotherapy history, hemoptysis, myocardial infarction or cerebrovascular accident within three months;
4. uncontrolled or active pulmonary inflammation;
5. participated in other clinical trials;
6. Pregnant women.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Estimated)
Dates: Start 2024-01-01 (Actual); Primary Completion 2026-01-01 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
2-year progression-free survival (PFS) | From the first day of radiotherapy to the occurrence of objective tumor progression or death due to any cause, whichever occurs first, assessed up to 60 months

SECONDARY OUTCOMES:
Overall Survival(OS) | From the first day of radiotherapy to the occurrence of death due to any cause, assessed up to 60 months
Local regional recurrence (LR) | From the first day of radiotherapy to the occurrence of clinical and/or biopsy-proven recurrence within the bronchial stump, ipsilateral hilum, mediastinum, or supraclavicular, whichever occurs first, assessed up to 60 months
Distant metastasis (DM) | From the first day of radiotherapy to the occurrence of any evidence of metastatic disease beyond the locoregional regions previously mentioned, assessed up to 60 months
Acute toxicity | From the first day of radiotherapy and up to the 3-month post-radiotherapy follow-up visit

CONTACTS AND LOCATIONS:
Overall Officials: jianyang wang, Principal Investigator — National Cancer Center
Locations (1):
- Department of Radiation Oncology,Cancer Institute and Hospital,Chinese, Beijing, Beijing Municipality, China

REFERENCES:
- [Background] Simon R. Optimal two-stage designs for phase II clinical trials. Control Clin Trials. 1989 Mar;10(1):1-10. doi: 10.1016/0197-2456(89)90015-9. PMID 2702835
- [Background] Jabbour SK, Lee KH, Frost N, Breder V, Kowalski DM, Pollock T, Levchenko E, Reguart N, Martinez-Marti A, Houghton B, Paoli JB, Safina S, Park K, Komiya T, Sanford A, Boolell V, Liu H, Samkari A, Keller SM, Reck M. Pembrolizumab Plus Concurrent Chemoradiation Therapy in Patients With Unresectable, Locally Advanced, Stage III Non-Small Cell Lung Cancer: The Phase 2 KEYNOTE-799 Nonrandomized Trial. JAMA Oncol. 2021 Jun 4;7(9):1-9. doi: 10.1001/jamaoncol.2021.2301. Online ahead of print. PMID 34086039
- [Background] Antonia SJ, Villegas A, Daniel D, Vicente D, Murakami S, Hui R, Kurata T, Chiappori A, Lee KH, de Wit M, Cho BC, Bourhaba M, Quantin X, Tokito T, Mekhail T, Planchard D, Kim YC, Karapetis CS, Hiret S, Ostoros G, Kubota K, Gray JE, Paz-Ares L, de Castro Carpeno J, Faivre-Finn C, Reck M, Vansteenkiste J, Spigel DR, Wadsworth C, Melillo G, Taboada M, Dennis PA, Ozguroglu M; PACIFIC Investigators. Overall Survival with Durvalumab after Chemoradiotherapy in Stage III NSCLC. N Engl J Med. 2018 Dec 13;379(24):2342-2350. doi: 10.1056/NEJMoa1809697. Epub 2018 Sep 25. PMID 30280658
- [Background] Zhou Q, Chen M, Jiang O, Pan Y, Hu D, Lin Q, Wu G, Cui J, Chang J, Cheng Y, Huang C, Liu A, Yang N, Gong Y, Zhu C, Ma Z, Fang J, Chen G, Zhao J, Shi A, Lin Y, Li G, Liu Y, Wang D, Wu R, Xu X, Shi J, Liu Z, Cui N, Wang J, Wang Q, Zhang R, Yang J, Wu YL. Sugemalimab versus placebo after concurrent or sequential chemoradiotherapy in patients with locally advanced, unresectable, stage III non-small-cell lung cancer in China (GEMSTONE-301): interim results of a randomised, double-blind, multicentre, phase 3 trial. Lancet Oncol. 2022 Feb;23(2):209-219. doi: 10.1016/S1470-2045(21)00630-6. Epub 2022 Jan 14. PMID 35038429
- [Background] Garassino MC, Mazieres J, Reck M, Chouaid C, Bischoff H, Reinmuth N, Cove-Smith L, Mansy T, Cortinovis D, Migliorino MR, Delmonte A, Sanchez JG, Chara Velarde LE, Bernabe R, Paz-Ares L, Perez ID, Trunova N, Foroutanpour K, Faivre-Finn C. Durvalumab After Sequential Chemoradiotherapy in Stage III, Unresectable NSCLC: The Phase 2 PACIFIC-6 Trial. J Thorac Oncol. 2022 Dec;17(12):1415-1427. doi: 10.1016/j.jtho.2022.07.1148. Epub 2022 Aug 9. PMID 35961520
- [Background] Cox JD, Stetz J, Pajak TF. Toxicity criteria of the Radiation Therapy Oncology Group (RTOG) and the European Organization for Research and Treatment of Cancer (EORTC). Int J Radiat Oncol Biol Phys. 1995 Mar 30;31(5):1341-6. doi: 10.1016/0360-3016(95)00060-C. No abstract available. PMID 7713792
- [Background] Han B, Li K, Wang Q, Zhang L, Shi J, Wang Z, Cheng Y, He J, Shi Y, Zhao Y, Yu H, Zhao Y, Chen W, Luo Y, Wu L, Wang X, Pirker R, Nan K, Jin F, Dong J, Li B, Sun Y. Effect of Anlotinib as a Third-Line or Further Treatment on Overall Survival of Patients With Advanced Non-Small Cell Lung Cancer: The ALTER 0303 Phase 3 Randomized Clinical Trial. JAMA Oncol. 2018 Nov 1;4(11):1569-1575. doi: 10.1001/jamaoncol.2018.3039. PMID 30098152
- [Background] Wang D, Bi N, Zhang T, Zhou Z, Xiao Z, Liang J, Chen D, Hui Z, Lv J, Wang X, Wang X, Deng L, Wang W, Wang J, Wang C, Lu X, Xu K, Wu L, Xue W, Feng Q, Wang L. Comparison of efficacy and safety between simultaneous integrated boost intensity-modulated radiotherapy and conventional intensity-modulated radiotherapy in locally advanced non-small-cell lung cancer: a retrospective study. Radiat Oncol. 2019 Jun 13;14(1):106. doi: 10.1186/s13014-019-1259-3. PMID 31196118
- [Background] Sun P, Li Y, Li C, Ren K, Wang Y, Yang H, Jiang W, Zou L, Yang H, Zhou H, Li ZM. A phase II study of sintilimab, anlotinib, and pegaspargase sandwiched with radiotherapy as first-line therapy in patients with newly diagnosed, stage I-II extranodal natural-killer/T-cell lymphoma. Am J Hematol. 2023 Jul;98(7):1043-1051. doi: 10.1002/ajh.26922. Epub 2023 Apr 7. PMID 36970971
- [Background] Li PJ, Lai SZ, Jin T, Ying HJ, Chen YM, Zhang P, Hang QQ, Deng H, Wang L, Feng JG, Chen XZ, Guo P, Chen M, Tian Y, Chen YY. Radiotherapy opens the blood-brain barrier and synergizes with anlotinib in treating glioblastoma. Radiother Oncol. 2023 Jun;183:109633. doi: 10.1016/j.radonc.2023.109633. Epub 2023 Mar 23. PMID 36963438
- [Background] He Z, Liu J, Ma Y, Jiang H, Cui Z, Wang G, Wu Y, Liu J, Cai X, Qian J, Huang J, Zhang H, Li H. Anlotinib Combined with Cranial Radiotherapy for Non-Small Cell Lung Cancer Patients with Brain Metastasis: A Retrospectively, Control Study. Cancer Manag Res. 2021 Aug 4;13:6101-6111. doi: 10.2147/CMAR.S319650. eCollection 2021. PMID 34377028
- [Background] Wozniak AJ, Moon J, Thomas CR Jr, Kelly K, Mack PC, Gaspar LE, Raben D, Fitzgerald TJ, Pandya KJ, Gandara DR. A Pilot Trial of Cisplatin/Etoposide/Radiotherapy Followed by Consolidation Docetaxel and the Combination of Bevacizumab (NSC-704865) in Patients With Inoperable Locally Advanced Stage III Non-Small-Cell Lung Cancer: SWOG S0533. Clin Lung Cancer. 2015 Sep;16(5):340-7. doi: 10.1016/j.cllc.2014.12.014. Epub 2015 Jan 9. PMID 25703100
- [Background] Lind JS, Senan S, Smit EF. Pulmonary toxicity after bevacizumab and concurrent thoracic radiotherapy observed in a phase I study for inoperable stage III non-small-cell lung cancer. J Clin Oncol. 2012 Mar 10;30(8):e104-8. doi: 10.1200/JCO.2011.38.4552. Epub 2012 Feb 13. No abstract available. PMID 22331948
- [Background] Spigel DR, Hainsworth JD, Yardley DA, Raefsky E, Patton J, Peacock N, Farley C, Burris HA 3rd, Greco FA. Tracheoesophageal fistula formation in patients with lung cancer treated with chemoradiation and bevacizumab. J Clin Oncol. 2010 Jan 1;28(1):43-8. doi: 10.1200/JCO.2009.24.7353. Epub 2009 Nov 9. PMID 19901100
- [Background] Auperin A, Le Pechoux C, Rolland E, Curran WJ, Furuse K, Fournel P, Belderbos J, Clamon G, Ulutin HC, Paulus R, Yamanaka T, Bozonnat MC, Uitterhoeve A, Wang X, Stewart L, Arriagada R, Burdett S, Pignon JP. Meta-analysis of concomitant versus sequential radiochemotherapy in locally advanced non-small-cell lung cancer. J Clin Oncol. 2010 May 1;28(13):2181-90. doi: 10.1200/JCO.2009.26.2543. Epub 2010 Mar 29. PMID 20351327
- [Background] O'Rourke N, Roque I Figuls M, Farre Bernado N, Macbeth F. Concurrent chemoradiotherapy in non-small cell lung cancer. Cochrane Database Syst Rev. 2010 Jun 16;2010(6):CD002140. doi: 10.1002/14651858.CD002140.pub3. PMID 20556756
- [Background] Bray F, Ferlay J, Soerjomataram I, Siegel RL, Torre LA, Jemal A. Global cancer statistics 2018: GLOBOCAN estimates of incidence and mortality worldwide for 36 cancers in 185 countries. CA Cancer J Clin. 2018 Nov;68(6):394-424. doi: 10.3322/caac.21492. Epub 2018 Sep 12. PMID 30207593